CLINICAL TRIAL: NCT00826254
Title: Nutritional Problems After Lung and Heart Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Foundation for Health and Rehabilitation (Other)
Responsible Party: Liv Forli, Rikshospitalet HF
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: S-03124 (REK); 2006/4716 (Personvernombud)
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2009-01

CONDITIONS: Bone Density; Overweight
Keywords: vitamin K; Bone Mineral Density; undercarboxylated osteocalcin
MeSH Terms: conditions — Overweight | interventions — Vitamin K; Soy Foods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Vitamin K — 180 micrograms vitamin K daily
  Other Names: Natto
Drug: Vitamin K — 2 capsules daily 180 micrograms vitamin K daily or placebo
  1 year
  Other Names: Natto

SUMMARY:
Part 1) Bone health after transplantation - possible influence of vitamin K

Part 2) Fat metabolism and endocrine parameters - possible predictors for developement of overweight after transplantation

ELIGIBILITY:
Inclusion Criteria:

* accepted for transplantation

Exclusion Criteria:

* not accepted for transplantation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2003-08; Primary Completion 2007-04 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
plasma vitamin K | 1 year

SECONDARY OUTCOMES:
Bone mineral density | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Liv Forli, Dr, Principal Investigator — Oslo University Hospital; Liv Forli, Dr, Study Director — Oslo University Hospital; Oystein Bjortuft, MD, Study Chair — Oslo University Hospital
Locations (1):
- Rikshospitalet HF, Oslo, Oslo County, Norway